CLINICAL TRIAL: NCT05916144
Title: The Effect of Interaction-Based Early Education Program Applied to Grandparents on the Growth and Development of Grandchildren
Brief Title: The Effect of Interaction-Based Early Education Program Applied to Grandparents on the Grandchildren's Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, mahmut caner us, Assoc Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09.2023.824
Record Dates: First submitted 2023-06-05; First posted 2023-06-23 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Grandparents; Growth Disorders; Development, Child; Feeding Behavior; Parent-Child Relations
Keywords: Grandparents; Grandchild; Growth and Development; Interaction Based Early Education Program; Parent-Child Relations
MeSH Terms: conditions — Growth Disorders; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The study was designed as a mixed methodology with semi-structured qualitative components for the pilot study and for post-intervention effectiveness while creating the intervention program, quantitative including pre-intervention and post-intervention analyses through scales.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and Outcome Assessors will be selected from medical students who did not have information about the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): The group in which grandparents actively participate in baby care, Grandparents with a score of 6 and above in the One Day of Life (Annex-5) questionnaire will be included.
  Interventions: Behavioral: Interaction-Based Early Education Program
- Group 2 (No Intervention): The group whose primary caregivers are mothers only

INTERVENTIONS:
Behavioral: Interaction-Based Early Education Program — The intervention program will be created based on the ETEÇOM model which is the Turkish adaptation of the Responsive Teaching Program developed in the United States. In this program, by improving the interactive behaviors of experts/educators or parents, the aim is for the child to acquire or develop 15 core behavior. Each session is planned to last between 60-90 minutes on average and will be conducted in a group format, consisting of 5 sessions, and can be conducted face-to-face or online.
  Arms: Group 1

SUMMARY:
In our study, "Does the early childhood intervention applied to grandparents as caregivers affect the child's growth, development (cognitive and socio-emotional development), and nutrition? Does early childhood intervention apply to grandparents as caregivers have an impact on caregiving characteristics, grandparent's health, attachment, parenting role, psychosocial well-being, role satisfaction, and communication with the child? Is early childhood intervention applied to grandparents as caregivers effective in creating a common language between grandparents and mothers on child care issues?" the answers to these questions will be tried to be answered.

This randomized controlled study will be conducted between July 2023 and July 2024 with children aged 0-4 years and their parents/grandparents using a mixed methodology. Children between the ages of 0-4 will be included in the study group, and those who are only cared for by their grandparents will be included in the study group, and cared for by their parents will be included in the control group.

The study will consist of 2 stages. The first phase will be conducted with a pilot study group to establish the training program. After the 5-session program is administered, a qualitative analysis will be made and the program will be finalized according to the feedback.

In the second stage of the study, a pre-test will be done through questionnaires, and then a training program will be applied to the group with grandparents as caregivers. The post-test will be applied to each group 6-8 weeks after the 5-group session ends. Pre-test and post-tests will be created in the online Google survey format. Pre-tests will only be applied to grandparents and mothers. Post-tests will be carried out at 4 practice times (after 6-8 weeks, 6th, 9th, and 12th months after the end of the intervention) determined for the evaluation of both parental and childhood outcomes. The second qualitative analysis will be made in a group format with the grandparents who applied for the program and the mothers (parents) of those children. For the qualitative analysis, the pre-created semi-structured interview format will be used after obtaining the consent of the participants, and if they give their consent, a voice recording will be taken. Fathers will also be informed and encouraged to participate and will be included in the qualitative phase of the study if they give consent for participation.

DETAILED DESCRIPTION:
Although the main focus in early childhood interventions is mother-child interaction, it is known that grandmothers are also culturally potential final decision makers in child care, especially in low- and low-middle-income countries (1). Therefore, given its role in child care, it has been emphasized that early childhood programs should offer a family-centred approach to child health by involving all key actors, including parents and grandmothers.

While studies have shown that the health of grandparents' grandchildren, and taking care of grandchildren from another point of view, have a mutual effect on the health of grandparents, it is also emphasized that more research needs to be done on this subject. In our study, "Does the early childhood intervention applied to grandparents as caregivers have an effect on the child's growth, development (cognitive and socio-emotional development), and nutrition? Does early childhood intervention apply to grandparents as caregivers have an impact on caregiving characteristics, grandparent's health, attachment, parenting role, psychosocial well-being, role satisfaction, and communication with the child? Is early childhood intervention applied to grandparents as caregivers effective in creating a common language between grandparents and mothers on child care issues?" The answers to the questions will be tried to be answered.

This is a randomized controlled study to be conducted between July 2023 and July 2024 with children aged 0-4 years and their parents/grandparents using mixed methodology. Children between the ages of 0-4 will be included in the study group, and those who are only cared for by their parents will be included in the control group. The study was designed as a mixed methodology with semi-structured qualitative components for the pilot study and for post-intervention effectiveness while creating the intervention program, quantitative including pre-intervention and post-intervention analyses through scales.

The study announcement will be announced on both posters and social media, and those who meet the inclusion criteria will be included in the study. The study will consist of 2 stages. The first phase will be carried out with a pilot study group to establish the training program. After the 5-session program is created on the basis of ETEÇOM, a qualitative analysis will be made and the program will be finalized according to the feedback.

In the second stage of the study, participants who meet the inclusion criteria will be randomly distributed to both groups until they reach the minimum number determined at the time of application, 10% more than the minimum number. Before each group, a pre-test will be done through questionnaires, a training program will be applied to the group with grandparents as caregivers, and the post-test will be applied to each group 6-8 weeks after the end. Pre-test and post-tests will be created in the online Google survey format. Pre-tests will only be applied to grandparents and mothers. Post-tests will be carried out at 4 practice times determined for the evaluation of both parental and childhood outcomes. In the last part of the study, qualitative analyzes will be made in a group format with the grandparents who applied for the program and the mothers (parents) of those children, and the study will be concluded. For the qualitative analysis, the pre-created semi-structured interview format will be used after obtaining the consent of the participants, and if they give their consent, a voice recording will be taken. Fathers will also be informed and encouraged to participate and will be included in the qualitative phase of the study if they give consent for participation.

Childhood outcomes will be evaluated in a total of 5 assessment periods. The first evaluation is the pretest, and after the second quantitative and in-depth qualitative analyzes are performed 6-8 weeks after the end of the intervention, the childhood outcomes will be re-evaluated in the 6th, 9th, and 12th months (3rd, 4th, and 5th quantitative tests) after the intervention. The first-year outputs will be taken as the basis for the thesis data, and it is planned to follow the study outputs until the 48th month.

Considering similar studies, it was planned to include at least 30 people in each group (20).

1. Group 1: The group in which grandparents actively participate in baby care, Grandparents with a score of 6 and above in the One Day of Life (Annex-5) questionnaire will be included in this group.
2. Group 2: The group whose primary caregivers are mothers only

ELIGIBILITY:
Inclusion Criteria:

Grandparents who have attended child care more than 2 times a week for at least 2 weeks and are known to continue to provide care support; Grandparents with grandchildren aged 0-4 who score 6 or higher on the "day of life" questionnaire will be included in the study group.

The control group will consist of mothers who are the primary caregivers of healthy children aged 0-4.

* Volunteer grandparents and mothers to be included in the study must be between the ages of 18-70.
* Participants are required to know, understand and speak Turkish fluently.

Exclusion Criteria:

* Known to have neurological and/or developmental problems, with chronic disease,
* 4 years or older or
* Those who refuse to participate in the study themselves or their families will be excluded from the study.

Ages: 1 Day to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The effect of the program on progress in Grandchild's socio-emotional and behavioural development by using the Brief Infant Toddler Social Emotional Assessment tool | 12 month after intervention
  The change from baseline in Brief Infant Toddler Social Emotional Assessment (BITSEA)problem subscale scores of grandchildren after the Responsive Teaching Program applied to caregiver Grandparents.
  BITSEA is a 42-item tool with 2 sub-scales: Problem (BITSEAP) and Competence (BITSEAc). Each item is scored as 0-1-2, with a maximum of 84 points and a minimum of 0 points. Higher total scores on BITSEAp indicate higher behavioural and emotional problems and lower total scores on BITSEAc indicate lower competency.
The effect of the program on Grandchild's developmental progress by using the Age and Stage Questionnaire | 12 month after intervention
  The change from baseline in Age and Stage questionnaire scores of grandchildren after the Responsive Teaching Program applied to caregiver Grandparents.

SECONDARY OUTCOMES:
The effect of the program on Grandparent's role satisfaction by using the Parental Stress Scale | 12 month after intervention
  The change from baseline in the Parental Stress Scale scores of Grandparents after the Responsive Teaching Program applied. The Parental Stress Scale is a 5-point Likert-type scale consisting of 16 items. Scored with a maximum of 80 points with a minimum of 0, with high scores indicating parental stress

CONTACTS AND LOCATIONS:
Overall Officials: Perran Boran, Prof., Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD can be shared with an acceptable reason

REFERENCES:
- [Background] Chung EO, Hagaman A, LeMasters K, Andrabi N, Baranov V, Bates LM, Gallis JA, O'Donnell K, Rahman A, Sikander S, Turner EL, Maselko J. The contribution of grandmother involvement to child growth and development: an observational study in rural Pakistan. BMJ Glob Health. 2020 Aug;5(8):e002181. doi: 10.1136/bmjgh-2019-002181. PMID 32784209
- [Background] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614
- [Background] Farrow C. A comparison between the feeding practices of parents and grandparents. Eat Behav. 2014 Aug;15(3):339-42. doi: 10.1016/j.eatbeh.2014.04.006. Epub 2014 May 9. PMID 25064278
- [Background] Pulgaron ER, Marchante AN, Agosto Y, Lebron CN, Delamater AM. Grandparent involvement and children's health outcomes: The current state of the literature. Fam Syst Health. 2016 Sep;34(3):260-269. doi: 10.1037/fsh0000212. Epub 2016 Aug 8. PMID 27505069
- [Background] Tanskanen AO, Danielsbacka M, Hamalainen H, Sole-Auro A. Does Transition to Retirement Promote Grandchild Care? Evidence From Europe. Front Psychol. 2021 Sep 20;12:738117. doi: 10.3389/fpsyg.2021.738117. eCollection 2021. PMID 34616345